CLINICAL TRIAL: NCT05316753
Title: Comparison of Biphasic Truncated Exponential and Pulsed Waveforms for Cardioversion of Atrial Fibrillation-High Energy Escalation Strategy and Introduction to Manual Pressure Application
Brief Title: BTE and Pulsed Waveforms for Cardioversion of Atrial Fibrillation - Escalation Strategy and Manual Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University National Heart Hospital (Other)
Responsible Party: Principal Investigator, Elina Trendafilova, professor, University National Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniversityNationalHeartH 1
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: electrical cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Intervention Model Description: Randomized Interventional study, Alternating Assignment, Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Schiller Defigard HD- 7 - DGHD7 (Experimental): Device: Cardioversion with a pulsed biphasic waveform Cardioversion is performed by a pulsed biphasic (Multipulse Biowave®) waveform (Schiller Defigard HD- 7 - DGHD7, Schiller Medical, France) with adult pads (0-21-0003 Schiller) following an energy protocol of 3 consecutive shocks with escalating selected energy: 150J, 200J, 200J. The third shock is combined with MAP (Manual Pressure Application). The protocol is stopped at successfull cardioversion (sinus rhythm at 1 min post-shock), otherwise after the 3rd shock Other Name: DGHD7
  Interventions: Procedure: Cardioversion with a pulsed biphasic waveform
- LIFEPAK 15, Physio-Control - LP15 (Active Comparator): Device: Cardioversion with a biphasic truncated exponential waveform Cardioversion is performed by a biphasic truncated exponential waveform (LIFEPAK 15, Physio-Control Inc., Redmond, WA, USA) with recommended by the manufacturer adult pads (Redipak QUICK COMBO, Physio-Control) following an energy protocol of 3 consecutive shocks with escalating selected energy: 150J, 360J, 360J. The third shock is combined with MAP (Manual Pressure Application). The protocol is stopped at successfull cardioversion (sinus rhythm at 1 minute post-shock), otherwise after the 3rd shock.
  Other Name: LP15
  Interventions: Procedure: Cardioversion with a biphasic truncated exponential waveform

INTERVENTIONS:
Procedure: Cardioversion with a pulsed biphasic waveform — Cardioversion with a pulsed biphasic waveform
  Other Names: Schiller Defigard HD- 7 - DGHD7, Schiller Medical, France
  Arms: Schiller Defigard HD- 7 - DGHD7
Procedure: Cardioversion with a biphasic truncated exponential waveform — Cardioversion with a biphasic truncated exponential waveform
  Other Names: LIFEPAK 15 monitor/defibrillator 41577-000267
  Arms: LIFEPAK 15, Physio-Control - LP15

SUMMARY:
Background: A Danish study raised the question of the usefulness of escalating energy protocols compared to fixed high-energy protocols. Maximal energies are usually the final choice of the physicians. Some authors showed that decreasing impedance by manual pressure application (MPA) had a positive impact on cardioversion outcome. This is likely due to the impedance decrease linked to MPA.

Objective: This new clinical cardioversion study of atrial fibrillation (AF) patients aims to compare the efficacy and safety of a new high energy escalation strategy. The protocol combines high energy shocks at first shock, jumping to maximal defibrillator energy at second shock and finally complemented by MPA at third shock, if success is not reached using electric shocks only.

Experimental design: Patients will be recruited at the Intensive Cardiology Care Unit, Cardiology Clinic, National Cardiology Hospital (NCH), Sofia, Bulgaria. All eligible patients will sign a written informed consent prior to the cardioversion and will receive the standard hospital procedures during cardioversion.

AF patients will be alternatively randomized to cardioversion using one of the two defibrillators, following the strategy below:

DEFIGARD HD-7 arm: 3 consecutive shocks with escalating selected energy: 150J, 200J, 200J. The third shock is combined with MPA LIFEPAK15 arm: 3 consecutive shocks with escalating selected energy: 150J, 360J, 360J. The third shock is combined with MPA The statistical power analysis will consider a superiority comparison between the cumulative energy actually delivered by both defibrillators.

The secondary cardioversion efficacy outcome measures are: the cumulative success rate (measured at 1 minute post-shock), number of delivered shocks. Delivered energy will be measured during each shock with a dedicated pulse recording device (approved by the NCH Ethical Committee). Heart rhythm will be measured in continuously recorded peripheral ECG.

The secondary cardioversion safety outcome measures are: markers for myocardial necrosis (high sensitive troponin I, CK-MB) evaluated on blood samples taken before and 8-12 hours after cardioversion; ST-segment changes (post-shock - pre-shock) measured in lead II; Complications after cardioversion measured during 2 hours follow-up period in the ICCU - the presence of apnea, arrhythmias, bradycardia and the need for respective therapy at the discretion of attending physician.

DETAILED DESCRIPTION:
Background Commercially available defibrillators generate direct current (DC) shock with various waveforms using distinct technologies. These waveforms are suggested to have different efficacy and safety. Although the superiority of biphasic over monophasic waveforms is well established, the relative efficacy and safety of the available biphasic waveforms is not clear.

Various BTE waveforms apply different potential gradients on the thorax that might produce various defibrillation effects. Apart from efficacy, the most important aspect is the patient safety, considering that larger potential gradients in the myocardium lasting longer could potentially induce an electroporation and then a fibrillation. A frequently observed effect of electroporation are the post-shock ST-segment deviations in the surface ECG, representing the potential difference between the normal tissue and sustained depolarized critical mass of myocardium closest to the associated origin of the electrical current. Although ST-segment changes are an easily ignored phenomenon, occurring acutely and resolving during the first few minutes post-shock, their presence in a short-term basis can identify electroporation by dangerously high potential gradients, while the sustained ST-changes in a long-term basis can identify cases with myocardial injury. The most reliable marker of shock-induced myocardial injuries is the high sensitive cardiac Troponin I (hsTnI).

In a previous study Trendafilova et al. were compared fixed-high energy protocols (200J-200J-200J) delivered by two different defibrillation waveforms: Pulsed (BTE-PE) and High-energy BTE (BTE-HE). This study concluded on non-inferiority between devices. Cumulative energy, efficiency of the waveforms and safety (measured by High-sensitive Troponin) were not reaching significant difference for both waveforms. Delivered energy of the first efficient shock was significantly lower for BTE-PE and although BTE-PE delivered almost 28J lower energy after the whole procedure, significance could not be reached due to wide variance.

In a Danish study Schmidt et al. compared two cardioversion protocols - one is fixed-high energy (360J-360J-360J), the other is low energy escalating (125J-150J-200J). The overall efficacy of fixed-energy protocol was better than escalating. Safety is non significantly different. Schmidt et al. raised the question of the usefulness of escalating energy protocols compared to fixed high-energy protocols.

There is an ethical consideration to apply maximal energy shocks to all patients without considering patient individuality. Ramirez et al. remind that failed shocks might depend on other factors like transthoracic impedance. Lavignasse et al. found that cumulative energy setting differs with patient characteristics, having significant association with: AF duration, gender, BSA, LV TDD, valvular disease and chronic respiratory disease. Indeed, some authors (Voskoboinik et al. and Ramirez et al.) showed that decreasing impedance by manual pressure application (MPA) had a positive impact on cardioversion outcome.

On most defibrillators, increasing the energy level is leading to an increase of the voltage delivered to the patient. This voltage increase implies a current increase in the thorax of the patient. In fact, applying a force on the defibrillation pads or increasing shock voltage by increasing the energy setting would lead to increase the current in the thorax, associated with expectations for higher shock efficiency. MPA is performed by pressing on the pads using a non-connected pair of paddles in order to assure isolation of the practitioner from the patient during the shock.

Objective:

This new clinical cardioversion study of atrial fibrillation (AF) patients aims to compare the efficacy and safety of a new high energy escalation strategy. The protocol combines reasonably high energy shocks complemented by MPA when necessary.

Two biphasic defibrillators - a standard BTE-HE waveform (Lifepak 15, Physio Control) and a BTE-PE waveform (Defigard HD 7, Schiller Medical) with different maximal energy settings of 360J and 200J, respectively are compared.

The proposed high energy escalation strategy is based on the hypothesis that most of the patients do not implicitly require the maximal levels of energy for cardioversion. Thus patients who could be easily cardioverted are removed from the pool that would need a more aggressive treatment.

Methods:

Study population All patients admitted for elective cardioversion of atrial fibrillation in ICCU- NCH will be potentially eligible for the study. Informed consent will be obtained from all eligible patients prior to cardioversion. Patients declining to participate in the study will receive treatment according to the hospital protocol.

Cardiologists will check the eligibility of each patient following the detailed list of inclusion and exclusion criteria, based on the documented pre-treatment data.

Additionally, eligibility will be verified through pre-cardioversion medical exams (blood test within 24 hours before cardioversion): routine blood chemistry, glucose, creatinine, eGFR, K, Na; CK-MB, high sensitive troponin I measurements on the day of cardioversion.

Study design This will be a prospective randomized trial (alternating design) where eligible patients will be randomized to treatment with two different defibrillators. Following the order of patient admittance in ICCU-NCH, the attending cardiologist will assign the odd and even eligible patients to the defibrillators in arm 1 and arm 2, respectively. The cardiologist cannot control the order of patient admittance in ICCU-NCH. The alternative randomization design will equalize the number of subjects on each treatment. This study is not designed to control for sex, age, comorbidity, type of device used for cardioversion, cumulative energy delivered during shocks, number of shocks administered. Randomization is performed to limit these and any other confounding factors.

Patient preparation Patients will be consulted prior to cardioversion (CV) in a quiet setting. Any questions will be answered by the attending cardiologist. Patients will be asked to manually sign their informed consent for study participation before further preparations and data collection. If the patient declines to participate, then he/she will receive treatment according to the hospital protocol without data documentation, as further defined in the study.

Demographic data will be taken. Pre-treatment data will be read from the patient files: concomitant diseases; medications during the previous 7 days; Left atrium dimensions, left ventricle dimensions and volumes, ejection fraction by transthoracic echocardiography during index hospitalization; TEE will be performed for all patients before CV - presence of cardiac thrombus and spontaneous echo contrast will be checked; duration of index AF in days; European Heart Rhythm Association class score of symptoms from index AF; standard blood test will be documented.

Appropriate standard anticoagulation with unfractionated heparin (UFH) or acenocumarol or direct oral anticoagulants (DOAC) is required before and after the CV.

The anesthesia will be conducted by an anesthesiologist with slow intravenous injection of Propofol, adjusted individually to reach deep sedation (Cook' s scale points <7).

Cardioversion protocol:

The CV procedure is performed in ICCU by a cardiologist and anesthesiologist. Defibrillator pads are placed according to the user guides on the pads and respecting >40 cm distance between them. Standard self-adhesive defibrillation pads, recommended by specific defibrillator's manufacturer will be used.

Defibrillator use: The time-interval interval between consecutive shocks is 1 min; The energy of consecutive shocks follows pre-defined protocol; The protocol stops at successful cardioversion (sinus rhythm at 1 min post-shock), otherwise at the last shock of the protocol.

Data collection and Follow up:

* Defibrillator pulse recorder: The shock waveforms delivered by the studied defibrillators is recorded in real-time during the shock by a dedicated measurement device (Defimpulse recorder DR2) connected in the patient circuit. This allows accurate measurement of the delivered energy, which is the primary measured outcome. Additionally, currents, voltages, patient impedances at each shock can be also measured. The device is fully automatic and expert assistance is not need during the CV intervention. The use of the measurement device (Defimpulse recorder DR2) has been approved by the NCH Ethical Committee.
* Blood samples, standard ECG, blood pressure and heart rate at baseline.
* Continuous ECG in 3 peripheral leads is recorded during the whole CV procedure. ST deviation is measured on the first cardiac complex after 10 s post-shock in standard manner (0.080 seconds after J point) in lead II.
* Standard ECG is recorded in 5 min after CV; 24 h after CV; at discharge if the discharge day is different from 24 h after CV.
* Heart rate and blood pressure are measured 3 times after CV during follow-up in ICCU
* Follow-up period in ICCU (2 hours after CV): Potential complications after CV are recorded
* Follow-up period in the Cardiology Clinic (24 hours after CV): blood samples to analyze CK-MB and troponin (8 to 12 h after CV); Clinical exam with heart rate and blood pressure; ECG; Any complications before discharge.

Statistics:

For arm1 (BTE PE waveform), the expected efficacy is 50% at the first shock (150J), 80% at the second shock (200J) and 85% at the third shock (200J combined with MPA).

For arm2 (BTE HE waveform), the expected efficacy is 50% at the first shock (150J), 80% at the second shock (360J) and 85% at the third shock (360J combined with MPA).

Taking into account that BTE PE waveform typically delivers 180J for energy setting of 200J, the estimated cumulative energy at the end of the CV procedure is 258J (+/-120J) and 366J (+/-240J) for arm1 and arm2, respectively.

The statistical analysis is designed for a superiority comparison between the two defibrillation strategies in respect of their delivered cumulative energies hypothesizing similar cardioversion efficacy rate. It is estimated that a total of 94 patients (47 per arm) would allow to reach a statistical power of 80% in a superiority study design with one-sided type I error rate of 0.05.

Continuous variables will be expressed as mean value ± standard deviation or median values (inter-quartile range) and compared with Students t-test or equivalent non-parametric test, respectively. Categorical variables are expressed as percentages and compared using the Chi-square or Fisher's exact test . P<0.05 is considered statistically significant for all comparisons.

Ethics All patients will sign a written informed consent prior to the cardioversion and will receive the standard hospital procedures during cardioversion. Both defibrillators included in this study are approved for clinical use and both are used on a daily basis.

Data anonymization policy will be respected. In order to ensure the medical confidentiality, no information about the patient will be entered in the defibrillators. An identification number will be given to each patient by the dedicated measurement device (Defimpulse recorder DR2). This number and the recording data are properties of the principal investigator. Approval from the NCH Ethical Committee concerning energy strategy and the use of the Defimpulse recorder during the cardioversion intervention has been obtained.

ELIGIBILITY:
Inclusion criteria:

* Indications for elective cardioversion of atrial fibrillation
* Patients > 18 years old and:
* Symptomatic AFIB with a duration of less than 12 months and EHRA score 2-4
* Symptomatic first detected AFIB and EHRA score 2-4
* Persistent AFIB after successful causal therapy
* Rare recurrences of AFIB with long periods of sinus rhythm
* Impossibility to reach a sustained normal ventricular rate in AFIB

Exclusion Criteria:

* Patients with atrial flutter
* Spontaneous HR <60/min
* Digitalis intoxication
* Impossibility to maintain sinus rhythm irrespective to antiarrhythmic therapy and frequent cardioversions
* Conduction disturbances (without fascicular block and AV block 1 degree) in patients without pacemaker
* Asymptomatic patients with AFIB for > 1 year
* Thyroid dysfunction: euthyroid status of at least one month is required (TSH is measured).
* Thrombosis in cardiac cavities, assessment performed using Transesophageal echocardiography (TEE)
* Spontaneous echo contrast > 2 degree (TEE)
* Patients with planned cardiac operation in the next three months
* Patients with embolic event in the last three months
* Patients <18 years of age
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Defibrillator Efficacy | Delivered energy (Joules) will be measured during each shock with a dedicated pulse recording device
  The cumulative delivered energy by the consecutive defibrillation shocks during the successful cardioversion procedure.

SECONDARY OUTCOMES:
The cumulative success rate at 1 minute | Peripheral ECG will be continuously recorded during cardioversion and the presence of sinus rhythm will be read by a cardiologist at the first minute after each shock
  The cumulative success rate (at 1 minute) of the consecutive defibrillation shocks during the cardioversion procedure is defined as the conversion to sinus rhythm at 1 minute post shock.
Number of shocks | During the whole cardioversion procedure, each electrical shock delivered to the patient will be counted
  Number of shocks
Changes in hsTnI at 8-12 hours | the blood samples will be taken before cardioversion (on the same day) and after cardioversion (from 8 to 12 hours after the intervention)
  Changes in hsTnI before and after the cardioversion procedure
Changes in CK and CK-MB at 8-12 hours | the blood samples will be taken before cardioversion (on the same day) and after cardioversion (from 8 to 12 hours after the intervention)
  Changes in CK and CK-MB before and after the cardioversion procedure before and after the cardioversion procedure
The cumulative success rate (at 2 hours) of the consecutive defibrillation shocks during the cardioversion procedure | Peripheral ECG will be continuously recorded during cardioversion and the presence of sinus rhythm will be read by a cardiologist at two hours after each shock
  The cumulative success rate (at 2 hours) of the consecutive defibrillation shocks during the cardioversion procedure, is defined as the conversion to sinus rhythm at 2 hours after the last shock of the procedure.
The cumulative success rate (at 24 hours) of the consecutive defibrillation shocks during the cardioversion procedure | Peripheral ECG will be continuously recorded during cardioversion and the presence of sinus rhythm will be read by a cardiologist at twenty four hours after each shock
  The cumulative success rate (at 24 hours) of the consecutive defibrillation shocks during the cardioversion procedure, is defined as the conversion to sinus rhythm at 24 hours after the last shock of the procedure.
ST-segment changes after each defibrillation shock | ST-segment will be measured in the continuously recorded lead II 10 seconds after each defibrillation shock (0.080 seconds after J point in the first QRS at 10 seconds post-shock)
  ST-segment changes after each defibrillation shock

CONTACTS AND LOCATIONS:
Overall Officials: Elina G Trendafilova, MD, PhD, Principal Investigator — UniversityNationalHeartH, ICCU
Locations (1):
- University National Heart Hospital, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavignasse D, Trendafilova E, Dimitrova E, Krasteva V. Cardioversion of Atrial Fibrillation and Flutter: Comparative Study of Pulsed vs. Low Energy Biphasic Truncated Exponential Waveforms. J Atr Fibrillation. 2019 Oct 31;12(3):2172. doi: 10.4022/jafib.2172. eCollection 2019 Oct-Nov. PMID 32435331
- [Background] Coats AJS, Anker SD, Baumbach A, Alfieri O, von Bardeleben RS, Bauersachs J, Bax JJ, Boveda S, Celutkiene J, Cleland JG, Dagres N, Deneke T, Farmakis D, Filippatos G, Hausleiter J, Hindricks G, Jankowska EA, Lainscak M, Leclercq C, Lund LH, McDonagh T, Mehra MR, Metra M, Mewton N, Mueller C, Mullens W, Muneretto C, Obadia JF, Ponikowski P, Praz F, Rudolph V, Ruschitzka F, Vahanian A, Windecker S, Zamorano JL, Edvardsen T, Heidbuchel H, Seferovic PM, Prendergast B. The management of secondary mitral regurgitation in patients with heart failure: a joint position statement from the Heart Failure Association (HFA), European Association of Cardiovascular Imaging (EACVI), European Heart Rhythm Association (EHRA), and European Association of Percutaneous Cardiovascular Interventions (EAPCI) of the ESC. Eur Heart J. 2021 Mar 31;42(13):1254-1269. doi: 10.1093/eurheartj/ehab086. PMID 33734354
- [Background] Ramirez FD, Sadek MM, Boileau I, Cleland M, Nery PB, Nair GM, Redpath CJ, Green MS, Davis DR, Charron K, Henne J, Zakutney T, Beanlands RSB, Hibbert B, Wells GA, Birnie DH. Evaluation of a novel cardioversion intervention for atrial fibrillation: the Ottawa AF cardioversion protocol. Europace. 2019 May 1;21(5):708-715. doi: 10.1093/europace/euy285. PMID 30535367
- [Background] Schmidt AS, Lauridsen KG, Torp P, Bach LF, Rickers H, Lofgren B. Maximum-fixed energy shocks for cardioverting atrial fibrillation. Eur Heart J. 2020 Feb 1;41(5):626-631. doi: 10.1093/eurheartj/ehz585. PMID 31504412
- [Background] Trendafilova E, Dimitrova E, Didon JP, Krasteva V. A Randomized Comparison of Delivered Energy in Cardioversion of Atrial Fibrillation: Biphasic Truncated Exponential Versus Pulsed Biphasic Waveforms. Diagnostics (Basel). 2021 Jun 17;11(6):1107. doi: 10.3390/diagnostics11061107. PMID 34204498
- [Background] Voskoboinik A, Moskovitch J, Plunkett G, Bloom J, Wong G, Nalliah C, Prabhu S, Sugumar H, Paramasweran R, McLellan A, Ling LH, Goh CY, Noaman S, Fernando H, Wong M, Taylor AJ, Kalman JM, Kistler PM. Cardioversion of atrial fibrillation in obese patients: Results from the Cardioversion-BMI randomized controlled trial. J Cardiovasc Electrophysiol. 2019 Feb;30(2):155-161. doi: 10.1111/jce.13786. Epub 2018 Nov 14. PMID 30375104